CLINICAL TRIAL: NCT04756102
Title: Early Pregnancy Glycemic Levels in Non-diabetic Primigravid Women and Pregnancy Outcome; Retrospective Study
Brief Title: Glucose Levels in Early Pregnancy and Feto-maternal Outcome
Status: Completed | Type: Observational
Sponsor: University of Jordan (Other)
Responsible Party: Principal Investigator, Naser Al-Husban, Assistant Professor, Jordan University Hospital
Other Study IDs: the University Of Jordan, Glu
Record Dates: First submitted 2021-02-08; First posted 2021-02-16 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2021-02

CONDITIONS: Maternal Diabetes
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- FBS lower than 80: Those pregnant patients with FBS less than 80 mg/dl
  Interventions: Other: Observation of their fetomaternal outcome
- FBS 80-120: Those pregnant patients with FBS between 80-120
  Interventions: Other: Observation of their fetomaternal outcome

INTERVENTIONS:
Other: Observation of their fetomaternal outcome — observe the fetal outcome and maternal outcome

SUMMARY:
to find out whether variations in the fasting blood glucose in early pregnancy affect the fetomaternal outcome

DETAILED DESCRIPTION:
Retrospective study conducted on the records of patients who were seen at Jordan University hospital in the period January 2016 to December 2020. All primigravid women with FBS that were done in early pregnancy before completed 20 weeks of gestation were included. Exclusion criteria were known diabetics, multiple pregnancies, thyroid dysfunction, patients taking steroids or any other medications for chronic illness (s) and those with missing data. Patients were divided into 2 groups; group had a FBS 80-120 mg/dl and group 2 with FBS less than 80 mg/dl. Pregnancy outcomes were then compared between the 2 groups.

Gestational age was confirmed by early ultra-sound (US) scan before 16 weeks gestation. All FBS samples were measured at our laboratory. Investigators collected data regarding patients' age, body mass index (BMI), FBS early in pregnancy, any complication in the pregnancy or the pregnancy outcome including miscarriage (defined as pregnancy loss before completed 24 weeks gestation), preterm delivery (defined as spontaneous vaginal delivery before completed 37 weeks gestation), gestational age at delivery, polyhydramnios, congenital abnormality (minor or major), stillbirth, intra-uterine fetal death (IUFD), neonatal death and mode of delivery. For those who underwent cesarean section, the indications were also identified. Fetal outcome included birth weight; APGAR score at 1 minute and APGAR score at 5 minutes. The APGAR score was determined by the neonatologists who routinely attend deliveries at our hospital.

Investigators also identified those who were diagnosed to have GDM with any intervention (metformin or insulin and their dosages). Diagnosis of GDM was based on a standard 75 gm glucose tolerance test (GTT) at 26-28 weeks gestation. A normal FBS level is lower than 95 mg/dL, one hour lower than 180 mg/dL, two hours lower than 155 mg/dL Three hours after drinking the glucose solution, a normal blood glucose level is lower than 140 mg/dL.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant

Exclusion Criteria:

* Thyroid disorder
* Diabetes mellitus
* Taking Steroids

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant women
Study Population: Pregnant women in their first pregnancy
Sampling Method: Non-Probability Sample
Enrollment: 218 (Actual)
Dates: Start 2018-01-30 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-12-15 (Actual)

PRIMARY OUTCOMES:
diagnosis of gestational diabetes | During her pregnancy; an average 20 weeks
  if the pregnant patients was diagnosed to have GDM

CONTACTS AND LOCATIONS:
Locations (1):
- Al-Husban University Naser, Amman, Jordan

IPD SHARING:
Plan to Share IPD: No